CLINICAL TRIAL: NCT03056547
Title: Biomarkers in Dyspnea
Acronym: BIODYSPNEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ADOREPS_5
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induced dyspnea (Experimental)
  Interventions: Other: Induced dyspnea

INTERVENTIONS:
Other: Induced dyspnea — Biological samples will be assessed during and after breathing discomfort induced by laboratory models of dyspnea ("work/effort", "air hunger").

SUMMARY:
To explore biological mechanisms in human model of induced dyspnea, in order to remove the source of dyspnoea, to modify cerebral impact and to allow the development of targeted therapies.

DETAILED DESCRIPTION:
The aim of the study will be to identify a specific biology and immunology associated with dyspnoea. It will open therapeutic possibilities through a better understanding of the mechanisms of dyspnea.

Healthy volunteers will underwent two types of dyspnea. The subjects will be first familiar with both types of dyspnea and dyspnea measurement scales. Different components of dyspnea will be measured.

Blood tests will be performed at different times (before dyspnea, during dyspnea, 60 and 90 min after dyspnea)

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy
* ongoing pain
* respiratory disease
* high levels of depression, panic disorder, or other significant mental health problems
* not fluent in french

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Biomakers in dyspnea | 60 minutes
  Biomarkers in human model of induced dyspnea

SECONDARY OUTCOMES:
Correlation with dyspnea intensity | 60 minutes
  Correlation between intensity of dyspnea and biomarkers
Correlation with dyspnea type | 60 minutes
  Correlation between type of dyspnea and biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique Paris Est - Groupe Hospitalier Pitié-Salpêtrière, Paris, France